CLINICAL TRIAL: NCT04816474
Title: The Effect of Training on Disease Management and Phone Counseling Service for Older Patients With Osteoarthritis on Functional Status, Self-Efficacy and Quality of Life
Brief Title: The Effects of Disease Management Training and Telephone Counseling Service for Elderly Patients With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: KTO Karatay University Evre
Record Dates: First submitted 2021-03-11; First posted 2021-03-25 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-02

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; nurse; self-efficacy; quality of life; functional status
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education and Phone Counseling Service (Experimental): Patients in this group will be trained online for 6 weeks. After the online training is over, a telephone consultation service will be provided once a week for 6 weeks.
  Interventions: Behavioral: Online education and Phone Counseling Service
- Control (No Intervention): No application will be made to patients in this group for 12 weeks. Pre-test and post-test will be applied.

INTERVENTIONS:
Behavioral: Online education and Phone Counseling Service — Online education total of 6 times for 6 weeks. Phone Counseling Service total of 6 times for 6 weeks
  Arms: Education and Phone Counseling Service

SUMMARY:
The study will be conducted to determine the difference on functional status, self-efficacy, and quality of life between groups with and without telephone counseling and training on disease management for participants.

DETAILED DESCRIPTION:
When the literature is examined, in patients with osteoarthritis who receive face-to-face training and intermittent telephone counseling; It is observed that the level of self-efficacy, compliance with the disease and quality of life have increased. It is stated that face-to-face training and telephone counseling services provided to participants on disease management will increase the effectiveness of education and as a result; It is thought that participants may have positive outcomes such as expressing their problems more easily, feeling safer by communicating frequently, and developing methods of coping with nurse-patient cooperation. When the studies conducted in our country are examined, while there are studies examining the effect of non-pharmacological interventions such as acupressor, hot-cold application, exercise training, mud pack treatment in patients with osteoarthritis; No study was found in the elderly patient group in which education and telephone counseling were conducted. The results of the research are thought to be beneficial in managing the disease in addition to in addition to pharmacological treatment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65 and over
* OA was diagnosed by the physician according to the American College of Rheumatology (ARD) criteria,
* Being able to answer research questions
* Individuals who gave their oral and written consent to participate in the study were included.

Exclusion Criteria:

* Having a history of malignancy
* Those who score above 5 points from the Visual Analogue Scale
* With a neuro psychiatric illness
* Having vision and hearing problems
* Receiving intraarticular medication (steroid, chondramine, hyaluronic acid) in the last month
* Surgery applied to the knee joint in the last 3 months
* Having inflammation in the joints
* Have an open wound in the OA area
* Individuals with a diagnosed vascular disease will not be included.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in functional status at 6 weeks and 12. weeks. | [Baseline, 6 weeks and 12 weeks]
  After the training and counseling, the functional status scores of the patients are checked. The Western 45 Ontario and McMaster Universities Osteoarthritis Index (WOMAC) scale has undergone several revisions. WOMAC; It consists of three subgroups: pain during various positions and movements, severity of joint stiffness, and difficulty in performing daily life activities. A total of 24 questions (pain 5, joint stiffness 2, physical function 17) and 5-point likert. In the evaluation, the questions are scored between 0 and 4 according to the Likert scale. The first option "no pain" is calculated as 0 points, the last option "very severe pain" is calculated as 4 points. Maximum scores of subgroups; 20 for pain, 8 for joint stiffness and 68 for physical function. The total score for each subgroup is the sum of the scores given to each item. As the scores get higher, symptoms worsen, restriction increases, and general health deteriorates.

SECONDARY OUTCOMES:
Change from baseline in self-efficacy at 6 weeks and 12. weeks. | [Baseline, 6 weeks and 12 weeks]
  After the interventions, the patient's self-efficacy scores are checked. Self-Efficacy Scale in Arthritis; It consists of 20 expressions evaluated on a visual scale with 10 digits, whose starting point is "I'm not sure = 1" and the other end is "I'm very sure = 10". It has four sub-dimensions: self-efficacy pain, self-efficacy hand and arm functions, self-efficacy foot leg functions and self-efficacy other symptoms. The first five statements are included in the self-efficacy pain sub-dimension and determine the level of pain coping in arthritis patients. The next nine statements are named self-efficacy hand-arm functions and self-efficacy foot leg functions, and are the two sub-dimensions of self-efficacy functions in the original. The minimum score of the scale is 20 and the maximum score is 200, and the higher the score is the indicator of the higher self-efficacy level.

OTHER OUTCOMES:
Change from baseline in life quality at 6 weeks and 12. weeks. | [Baseline, 6 weeks and 12 weeks]
  After the interventions, the patient's life quality scores are checked. The World Health Organization Quality of Life Scale Elderly Module, the older module of World Health Organization Quality of Life Scale, Bullinger et al. developed by. The World Health Organization Quality of Life Scale Elderly Module consists of 24 questions in six dimensions where the answers are determined with a five-point Likert scale. These six dimensions are: "sensory functions" (questions 1, 2, 10 and 20), "Autonomy" (questions 3, 4, 5 and 11), "Past, Present, Future Activities" (12, 13, 15). and questions 19), "Social participation" (questions 14,16, 17 and 18), "death and dying" (questions 6, 7, 8 and 9) and "Intimacy" (questions 21, 22, 23 and 24). questions). Possible dimension scores range from 4-20. Also, the "total score" can be calculated by adding up the individual point values. The higher the score, the better the quality of life.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Akademi Hastanesi, Konya
  - Konya Meram Akademi Hastanesi, Konya

IPD SHARING:
Plan to Share IPD: No
After the research is completed.

REFERENCES:
- [Derived] Yilmaz E, Polat U. Online Disease Management Training for Older Adults With Osteoarthritis: A Randomized Controlled Trial. Musculoskeletal Care. 2024 Sep;22(3):e1931. doi: 10.1002/msc.1931. PMID 39134868